CLINICAL TRIAL: NCT00575497
Title: Study of Clinical Outcomes of More Frequent Hemodialysis
Brief Title: More Frequent Dialysis (>3 Treatments Per Week)
Acronym: MFD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SR002MFD
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: End Stage Renal Disease; Chronic Kidney Disease
Keywords: Hemodialysis; Adequacy; Frequency
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- A (Experimental): Six Day per week short daily hemodialysis
  Interventions: Procedure: More frequent hemodialysis
- B (Experimental): Six nights per week nocturnal hemodialysis
  Interventions: Procedure: More frequent hemodialysis
- C (Experimental): Every other day short daily hemodialysis
  Interventions: Procedure: More frequent hemodialysis
- D (Experimental): Every other night hemodialysis
  Interventions: Procedure: More frequent hemodialysis
- E (Experimental): 5 days per week short daily hemodialysis
  Interventions: Procedure: More frequent hemodialysis
- F (Experimental): 5 nights per week hemodialysis
  Interventions: Procedure: More frequent hemodialysis
- G (Active Comparator): Conventional three time per week short daily hemodialysis
  Interventions: Procedure: Conventional Hemodialysis

INTERVENTIONS:
Procedure: More frequent hemodialysis — Six Day per week short daily hemodialysis
  Arms: A
Procedure: More frequent hemodialysis — Six nights per week nocturnal hemodialysis
  Arms: B
Procedure: More frequent hemodialysis — Every other day short daily hemodialysis
  Arms: C
Procedure: More frequent hemodialysis — Every other night hemodialysis
  Arms: D
Procedure: More frequent hemodialysis — 5 days per week short daily hemodialysis
  Arms: E
Procedure: More frequent hemodialysis — 5 nights per week hemodialysis
  Arms: F
Procedure: Conventional Hemodialysis — 3 days per week short daily hemodialysis
  Arms: G

SUMMARY:
The study compares the benefits of short daily hemodialysis six days a week, nocturnal (night time) hemodialysis six days a week, every other day and every other night hemodialysis to traditional three days a week hemodialysis.The hypothesis is that increasing hemodialysis treatment time and/or frequency will improve outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Stable vascular access, i.e., lack of needling difficulties and stable flow rates. Accesses will include fistulae, grafts, catheters and ports.
* 18 years of age.
* History of compliance with a dialysis treatment schedule, or if a new patient, express a willingness to be compliant with a treatment schedule.
* Plan to continue care and follow-up at the investigational site.
* Able to sign the informed consent and other relevant documents.

Exclusion Criteria:

* History of poor compliance with thrice (or twice) weekly dialysis schedules as manifested by more than three unexplained missed treatments in the past six (6) months.
* Pregnancy.
* Intravenous drug abuser.
* Expects to receive a transplant or transfer to another facility within six months of entering the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2005-01; Primary Completion 2012-08-07 (Actual); Study Completion 2012-08-07 (Actual)

PRIMARY OUTCOMES:
Hospitalization days per year | Ongoing

SECONDARY OUTCOMES:
Nutritional Status measured by Subjective Global Assessment | Ongoing
Anemia, measured by erythropoetin dose | Ongoing
Control of hypertension, as measured by number of antihypertensive tablets taken per day | Ongoing
Control of hyperphosphatemia, as measured by number of phosphate binder tablets taken per day | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: John Moran, MD, Study Director — Satellite Healthcare, Inc.; Brigittte Schiller-Moran, MD, Principal Investigator — Satellite Healthcare, Inc.
Locations (2):
- United States (2):
  - Satellite Healthcare, Inc., Mountain View, California
  - WellBound, Inc., Mountain View, California